CLINICAL TRIAL: NCT04894214
Title: Flow-controlled Ventilation (FCV) in Moderate Acute Respiratory Distress Syndrome (ARDS) Due to COVID-19 - an Interventional Cross-over Study
Brief Title: Flow-controlled Ventilation (FCV) in Moderate Acute Respiratory Distress Syndrome (ARDS) Due to COVID-19
Acronym: VICAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, Principal investigator, Member of staff at the department of critical care, Doctor of Philosophy, Medical Doctor, University Hospital, Antwerp
Other Study IDs: 001533; 001533 (Other: EDGE)
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Respiration, Artificial
Keywords: Flow controlled ventilation (FCV)
MeSH Terms: conditions — Respiratory Aspiration | interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Point-of-care arterial blood gas sampling. The sample will be disposed as biohazard material after analysis is done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sequential "baseline PCV" - "FCV" - "VCV": Each participant will be subjected to baseline pressure controlled ventilation (PCV) during 5 minutes, followed by 30 minutes of FCV with an evone respirator (Ventinova Medical B.V., Eindhoven, The Netherlands) and eventually 30 minutes of VCV. Respiratory rate (RR), positive end-expiratory pressure (PEEP) and inspiratory fraction of oxygen (FiO2) will be held constant. According to the manufacturers guidelines, an I:E ratio of 1:1 will be pursued during FCV. During FCV, the respirator will be set with the same PIP as during baseline PCV. For VCV, the same tidal volume as during baseline PCV will be set.
  Interventions: Diagnostic Test: Arterial blood gas (ABG); Other: Recording of hemodynamic monitoring; Other: Recording of respiratory monitoring

INTERVENTIONS:
Diagnostic Test: Arterial blood gas (ABG) — Arterial blood gasses will be drawn during baseline PCV, and every 15 minutes during FCV and VCV respectively. pO2 (mmHg), pCO2 (mmHg) and pH will be recorded.
Other: Recording of hemodynamic monitoring — Hemodynamic parameters (invasive arterial blood pressure (mmHg) and heart rate (beats per minute)) will be recorded every 5 minutes.
Other: Recording of respiratory monitoring — Tidal volume (ml), respiratory rate (breaths per minute), minute volume (l/min), dynamic compliance (ml/cmH2O), resistance (cmH2O/l/min), plateau pressure (cmH2O), mean airway pressure (cmH2O), positive end-expiratory pressure (cmH2O), peak inspiratory pressure (cmH2O) and fraction of inspired oxygen will be recorded every 5 minutes.

SUMMARY:
Flow controlled ventilation (FCV) is a fairly new mode of mechanical ventilation, consisting of a constant inspiratory and expiratory flow. Inspiration is thus comparable to volume controlled ventilation (VCV). The actively controlled, constant flow during expiration is unique. FCV is known to minimize dissipated energy to the lung [ref] and is therefore supposed to aid in lung protective ventilation.

The VICAR study is designed as a prospective single cohort crossover trial. The intervention consists of a sequence of respiratory modes: baseline pressure controlled ventilation (PCV) during 5 minutes, followed by 30 minutes of FCV with an evone respirator (Ventinova Medical B.V., Eindhoven, The Netherlands) and eventually 30 minutes of VCV. Every participant will receive the intervention. Respiratory rate (RR), positive end-expiratory pressure (PEEP) and inspiratory fraction of oxygen (FiO2) will be held constant. According to the manufacturers guidelines, an I:E ratio of 1:1 will be pursued during FCV. During FCV, the respirator will be set with the same PIP as during baseline PCV. For VCV, the same tidal volume as during baseline PCV will be set.

ELIGIBILITY:
Inclusion Criteria:

* P/F-ratio: 100-200 (moderate ARDS)
* SpO2 88-94%
* PaO2 60-80 mmHg
* COVID-19 positive on a PCR test

Exclusion Criteria:

* BMI > 40 kg/m²
* Prone ventilation
* Already invasively mechanically ventilated for more than 10 days
* Refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring mechanical ventilation for moderately severe ARDS (P/F ratio 100-200) due to COVID-19 were recruited from a tertiary intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen tension, PaO2 (mmHg) | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Arterial partial oxygen tension as measured on an arterial blood gas sample.
P/F ratio or Horowitz index (mmHg) | Post hoc calculation
  Ratio of the arterial oxygen tension PaO2 (mmHg) divided by the inspiratory fraction of oxygen FiO2.

SECONDARY OUTCOMES:
SpO2 (%) | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Oxygen saturation as measured by pulse oxymetry.
FiO2 | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Fraction of inspired oxygen as measured by the respirator.
PEEP (cmH2O) | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Positive end-expiratory pressure as measured by the respirator.
Pmean | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Mean airway pressure (cmH2O) as measured by the respirator.
PaCO2 | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Arterial partial tension of carbon dioxide (mmHg) as measured on an arterial blood gas sample.
MV | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Minute volume (l/min) as measured by the respirator.
TV | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Tidal volume (ml) as measured by the respirator.
RR | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Respiratory rate (breaths per minute) as measured by the respirator.
Pplat | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Plateau airway pressure (cmH2O) as measured by the respirator
PIP | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Peak inspiratory airway pressure (cmH2O) as measured by the respirator.
ABPsys | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Systolic arterial blood pressure (mmHg) as measured by a pressure transducer on an arterial catheter.
ABPmean | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Mean arterial blood pressure (mmHg) as measured by a pressure transducer on an arterial catheter.
ABPdia | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Diastolic arterial blood pressure (mmHg) as measured by a pressure transducer on an arterial catheter.
HR | Approximately 1 hour (5 min. PCV + 30min. FCV + 30 min. VCV)
  Heart rate (beats per minute) as measured on a 5-lead continuous electrocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Schepens, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van Dessel ED, De Meyer GR, Morrison SG, Jorens PG, Schepens T. Flow-controlled ventilation in moderate acute respiratory distress syndrome due to COVID-19: an open-label repeated-measures controlled trial. Intensive Care Med Exp. 2022 May 24;10(1):19. doi: 10.1186/s40635-022-00449-4. PMID 35608696